CLINICAL TRIAL: NCT06908252
Title: Integrating PrEP Into Mobile Addiction Treatment and Primary Care Services
Brief Title: MAPS PrEP Van Study
Acronym: MAPS PrEP
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: Pro00116108; 5P30AI064518-20 (NIH)
Record Dates: First submitted 2025-03-20; First posted 2025-04-03 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: HIV Infection
Keywords: People who inject drugs; Mobile Medical Unit; PrEP; Syringe Service Program; HIV prevention
MeSH Terms: conditions — HIV Infections | interventions — Pre-Exposure Prophylaxis

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- PrEP (Experimental): All eligible participants will be given oral PrEP pills to reduce their risk for contracting HIV.
  Interventions: Drug: Pre-Exposure Prophylaxis (PrEP)

INTERVENTIONS:
Drug: Pre-Exposure Prophylaxis (PrEP) — Oral Pre-Exposure Prophylaxis (PrEP) pills

SUMMARY:
For this study the investigators aim to see if giving participants an oral HIV prevention medication on a medical van, is a good option of care for individuals who inject drugs and/or are sexually active and therefore at a higher risk of contracting HIV.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate a pilot program that provides Pre-Exposure Prophylaxis (PrEP) for people who use drugs (PWUD) and are at risk for contracting HIV. Given the ongoing overdose crisis and the risk of HIV among PWUD, this study aims to assess weather offering oral PrEP on a Medical Mobile Unit (MMU) is a viable strategy for preventing HIV transmission in high-risk populations. The other goal of this study is to assess community perceptions of PrEP and perceived HIV risk among Syringe Service Program (SSP) clients visiting a MMU.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older, active drug injection user and/or sexually active, referred from the Syringe Service Program

Exclusion Criteria:

* positive HIV status

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-09-17 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Enrollment | Baseline
  Number of participants utilizing medical mobile unit during study duration who are eligible for PrEP
Negative HIV Status | up to 3 months
  Number of participants who remain HIV negative at 3 months (Measured via negative HIV test at 3 months
PrEP Consultation | up to 6 months
  Number of participants who agree to PrEP consultation
PrEP Initiation | up to 6 months
  Number of participants who complete PrEP consultation and start PrEP
Retention | up to 6 months
  Number of participants who come back for 3 month and 6 month visit
Follow Through | up to 6 months
  Number of participants who pick up PrEP medication
Negative HIV Status at 6 months | up to 6 months
  Number of participants who remain HIV negative at 6 months (Measured via negative HIV test at 6 months)

CONTACTS AND LOCATIONS:
Overall Officials: Mehri McKellar, MD, Principal Investigator — Duke Health; Jacqueline Hodges, MD, MPH, Principal Investigator — Duke Health
Locations (1):
- Duke Department of Population Health Sciences, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No